CLINICAL TRIAL: NCT02823340
Title: Fractionated Microneedle Radiofrequency for Treatment of Primary Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, xjpfW, chief of dermatology, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJPFMR-201506
Record Dates: First submitted 2016-06-16; First posted 2016-07-06 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Primary Axillary Hyperhidrosis

ARMS (1):
- Fractional Microneedle Radiofrequency Treatment (Experimental): Fractional Microneedle Radiofrequency Treatment
  Interventions: Device: Fractional microneedle RF(United, Peninsula Medical, China)

INTERVENTIONS:
Device: Fractional microneedle RF(United, Peninsula Medical, China)

SUMMARY:
Twenty patients with PAH had 1 session of Fractionated microneedle radiofrequency treatment. Clinical improvement was evaluated using a Hyperhidrosis Disease Severity Scale (HDSS) and photographs were taken using the starch-iodine test at every visit and 4 weeks, 8 weeks, and 24 weeks after the treatment. Skin biopsies were obtained from 3 of the enrolled patients before and after treatment. The satisfaction and adverse reactions of the research participants were recorded at every follow-up visit.

DETAILED DESCRIPTION:
Hyperhidrosis Disease Severity Scale (HDSS)Score = 1 My sweating is never noticeable and never interferes with my daily activitiesScore = 2 My sweating is tolerable but sometimes interferes with my daily activitiesScore = 3 My sweating is barely tolerable and frequently interferes with my daily activitiesScore = 4 My sweating is intolerable and always interferes with my daily activities

ELIGIBILITY:
Inclusion Criteria: Meet the following conditions

* Diagnosed according to having a score of 3 or 4 on a Hyperhidrosis Disease
* Severity Scale (HDSS);
* Patients aged 18 to 40 years (to the date of screening);
* Not treatment in Axillary area before;
* Understanding the whole process of the study, voluntary participation and signed the informed consent;
* Patient compliance is good, can guarantee in course of observation.

Exclusion Criteria:One of the following is not included in this study:

* Pregnant women, ready to pregnant or lactating women;
* Have a serious heart, lung, kidney and other vital organs and endocrine system lesions and the history
* Need insulin control of diabetes; High blood pressure did not get good controller ;
* Patients with white blood cells <4.0 × 109 / L, or a definite anemia (hemoglobin less than 100g / L), or platelets <100 × 109 / L, or other blood disease;
* Patients with chronic diarrhea, or peptic ulcer nearly 1 year;
* Patients suffering from malignant tumor;
* Patients suffering from acute and chronic infectious diseases;
* Mental disorders, history of alcohol abuse, drug or other substance abuse;
* Other cases which researchers believe that can not enroll.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The improvement of Hyperhidrosis Disease Severity Scale (HDSS) | up to 24 weeks

SECONDARY OUTCOMES:
The improvement of visual analog scale(VAS) by patient | 0 week, 4weeks, 8weeks, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospitial, Xi'an, Shaanxi, China